CLINICAL TRIAL: NCT05427279
Title: Investigating the Effects of 24-hours of Repeated Doses of Vitamin C Enriched Hydrolyzed Collagen, PrimaColl™, Whey Protein, or Placebo on Collagen Synthesis
Brief Title: Effects of Vitamin C Enriched Hydrolyzed Collagen, PrimaColl™, Whey Protein, or Placebo on Collagen Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Geltor (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 220518
Record Dates: First submitted 2022-06-09; First posted 2022-06-22 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Effect of Food Supplement
Keywords: Collagen synthesis; Exercise; Supplementation; Engineered ligaments
MeSH Terms: conditions — Motor Activity | interventions — maltodextrin; Whey Proteins

STUDY DESIGN:
Intervention Model Description: Participants will consume a supplemental dose of hydrolyzed collagen (20g with 50mg vitamin C), PrimaColl (20g with 50mg vitamin C), whey protein (20g whey isolate with 50mg vitamin C) or a placebo (20g maltodextrin with 50mg vitamin C) 1hr prior to exercise bouts (6 minutes of jump rope). The type of consumed supplementation will be randomized where neither the participant nor investigator will know which supplement is being consumed. Each participant will repeat the protocol four times.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which treatment. The interventions will be coded using a blinded alphabetical letter code (A, B, C, D). A delegate researcher (independent party not further involved in the study) will randomize all interventions using a computer-generated randomization list. The delegate will hand in the code-breaker to the principal investigator in a sealed envelope. The envelope will be stored in a locked filing cabinet in the principal investigator's office, which will also be locked when unoccupied. The envelope will be opened by the principal investigator after completing the analysis of blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): This arm will be given a placebo (20g maltodextrin with 50mg vitamin C)
  Interventions: Dietary Supplement: Placebo
- Hydrolized Collagen (Experimental): This arm will be given Hydrolized Collagen (20g with 50mg vitamin C)
  Interventions: Dietary Supplement: Hydrolized Collagen
- PrimaColl (Experimental): This arm will be given PrimaColl, a vegan collagen supplementation (20g with 50mg vitamin C)
  Interventions: Dietary Supplement: PrimaColl
- Whey Protein (Experimental): This arm will be given whey protein (20g with 50mg vitamin C)
  Interventions: Dietary Supplement: Whey protein

INTERVENTIONS:
Dietary Supplement: Placebo — The participant will consume a supplemental dose of a placebo (20g maltodextrin with 50mg vitamin C)
  Other Names: maltodextrin
  Arms: Placebo
Dietary Supplement: Hydrolized Collagen — The participant will consume a supplemental dose of Hydrolized collagen (20g with 50mg vitamin C)
  Arms: Hydrolized Collagen
Dietary Supplement: PrimaColl — The participant will consume a supplemental dose of PrimaColl, a vegan collagen supplementation (20g with 50mg vitamin C)
  Arms: PrimaColl
Dietary Supplement: Whey protein — The participant will consume a supplemental dose of whey protein (20g whey isolate with 50mg vitamin C)
  Arms: Whey Protein

SUMMARY:
The purpose of this study is to determine the effects of repeated dosing vitamin C enriched hydrolyzed collagen (HC) over a 24hr period, compared to PrimaColl™ (PC), whey protein (WP) and placebo (PL), with prescribed exercise on collagen synthesis.

To achieve this, participants will consume a supplemental dose of HC (20g with 50mg vitamin C), PC (20g with 50mg vitamin C), whey protein (20g whey isolate with 50mg vitamin C) or a placebo (20g maltodextrin with 50mg vitamin C) 1hr prior to an exercise bout (6 minutes of jump rope), this will be repeated three times over a 24h period.

The amount of collagen protein synthesized will be indirectly measured by measuring pro-collagen type I N-terminal propeptide (PINP) in the serum before and 4hrs after the last exercise bout.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of repeated dosing of vitamin C enriched hydrolyzed collagen (HC) over a 24hr period, compared to PrimaColl™ (PC), whey protein (WP) and placebo (PL), with prescribed exercise on collagen synthesis.

To achieve this, participants will consume a supplemental dose of HC (20g with 50mg vitamin C), PC (20g with 50mg vitamin C), whey protein (20g whey isolate with 50mg vitamin C) or a placebo (20g maltodextrin with 50mg vitamin C) 1hr prior to exercise bouts (6 minutes of jump rope). The amount of collagen protein synthesized will be indirectly measured by measuring procollagen type I N-terminal propeptide (PINP) in the serum before and 4hrs after the last exercise bout.

It is expected that this project will determine whether greater increases in collagen synthesis are observed with repeated doses of HC and exercise, compared with a single dose and exercise bout (from previous research). This study will also determine whether collagen synthesis is similarly stimulated with PrimaColl, or whey protein. Results from this study will help to better prescribe the use of dietary collagen and exercise training to improve collagen synthesis in healthy young people. Improved collagen synthesis has the potential to decrease ligament, tendon, and bone injuries in the general and athletic populations.

Male and female participants between the ages of 18-30 years of age will be enrolled in the study. A randomized double-blind crossover design with neither the subjects nor the investigators knowing who is on which treatment (HC, PC, WP or PL).

I. Baseline blood draw

The subjects will arrive in the laboratory following an overnight fast. The antecubital vein will be cannulated, and an initial 5 mL baseline blood sample will be collected.

II. Supplementation

After baseline blood draw subjects will be provided with a supplement as shown in the table below. Subjects will be asked to consume the supplement that will be pre-mixed with 250 ml of water 60 min before the jump rope exercise. This will be repeated 3 times, separated by 12 hours over a 24h period.

III. Exercise

Sixty minutes after the ingestion of the supplement, each participant will complete 6 minutes of jump rope. This will be repeated on 3 occasions over a 24hr period. Subjects will be asked to abstain from vigorous exercise during the 24hr period, aside from the prescribed jump rope exercise.

Subjects will be asked to ingest supplement and jump rope in lab for time point 1. Subjects will be given the option to ingest supplement and jump rope outside lab if more conducive to their scheduling restrictions at time points 2 and 3 blood draws are not required at these timepoints. Subjects will be asked to return to the lab 4 hours after last jumping session for blood sampling.

Blood draws for PNIP analysis

Blood samples (5 mL) at different time points:

* Baseline 2 vials will be drawn (1 for PINP and the other for bioassays)
* 1h after the first supplementation 1 vial will be drawn (bioassay)
* 4hrs post-exercise session number 3 the last vial will be drawn (PINP) Blood will be collected in 5 mL serum separating tubes and allowed to clot for 1hr before centrifugation at 1000 x g for 10 minutes and the serum will be frozen and kept at -30°C until processed. PINP levels will be determined by electrochemiluminescence (ECL; Roche Diagnostics, Indianapolis, IN) according to the manufacturer's instructions. The total number of blood draws will be 12 (3 per intervention with 4 interventions). Treatments will be randomized to avoid an order effect and a washout period of about 72h between trials will be used to minimize the effect of the previous treatment

ELIGIBILITY:
Inclusion Criteria:

* healthy active male or female
* normal weight (BMI between 18 and 25 kg/m2)

Exclusion Criteria:

* taking any medication that may interfere with the study
* have a history of more than 3 musculoskeletal injuries within the past 12 months
* have any health or dietary restriction that would be affected by the supplementation protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Collagen protein synthesis | Baseline (0 hour) to 4 hours after last exercise bout (at 28 hour of the protocol)
  Collagen protein synthesis will be indirectly measured by measuring pro-collagen type I N-terminal propeptide (PINP) in the serum before and 4 hours after the last exercise bout (at 28 hours of the protocol)

SECONDARY OUTCOMES:
Ligament collagen content | Baseline (0 hour) to directly after consumption of supplementation (1 hour)
  Serum from participants will be used to treat engineered ligaments in order to assess the effect of the different supplementation on the ligament collagen content using a hydroxyproline assay kit.
Strength of engineered ligaments | Baseline (0 hour) to directly after consumption of supplementation (1 hour)
  Serum from participants will be used to treat engineered ligaments in order to measure the effect of the different supplementation on the strength of the ligaments, the strength will be measured using the Instron bio puls 68SC-1 tension and compression machine.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Baar, PhD, Principal Investigator — UC Davis
Locations (1):
- Hickey Laboratory, Davis, California, United States